CLINICAL TRIAL: NCT03523338
Title: An Open-Label Expanded Access Protocol for Apalutamide Treatment of Subjects With Non Metastatic Castration-Resistant Prostate Cancer
Brief Title: An Expanded Access Protocol for Apalutamide Treatment of Participants With Non-Metastatic Castration-Resistant Prostate Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108434; 2017-004203-41 (EudraCT Number); 56021927PCR3010 (Other: Aragon Pharmaceuticals, Inc.)
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Androgen Antagonists; Standard of Care

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Apalutamide — Participants will receive apalutamide 240 mg orally once daily.
  Other Names: JNJ-56021927
Drug: ADT (Standard of Care) — Participants who did not undergo surgical castration, should receive and remain on a stable regimen of ADT according to local standard of care.

SUMMARY:
The purpose of this study is to collect additional safety data until apalutamide is commercially available for participants with non-metastatic castrate-resistant prostate cancer (NM-CRPC).

ELIGIBILITY:
Inclusion Criteria:

* Participants with confirmed prostate cancer, with evidence of castration resistance, with a rising prostate-specific antigen (PSA) while on androgen deprivation therapy (ADT), and for whom the treating physician believes additional therapy is indicated in the non-metastatic castrate-resistant prostate cancer (NM-CRPC) setting

  a) Willingness to continue gonadotropin releasing hormone analog (GnRHa) throughout study if the participant is medically castrated
* Must sign an informed consent form (ICF) (or the participant's legally acceptable representative must sign) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
* To avoid risk of drug exposure through the ejaculate (even participants with vasectomies), participants must use a condom during sexual activity while on study drug and for 3 months following the last dose of study drug. Donation of sperm is not allowed while on study drug and for 3 months following the last dose of study drug
* Willingness and ability to comply with prohibitions and restrictions specified in this protocol, scheduled visits, treatment plans, laboratory, and other study procedures, including ability to swallow study drug tablets

Exclusion Criteria:

* Previously enrolled in another apalutamide study or eligible for enrollment in another ongoing clinical study of apalutamide
* Enrolled in another interventional clinical study of anti-neoplastic agents
* Ongoing grade greater than (>) 1 acute toxicity due to prior therapy or surgical procedure
* Concurrent therapy with medications known to lower the seizure threshold must have been discontinued or substituted at least 4 weeks prior to study entry
* Current or prior treatment with anti-epileptic medications for the treatment of seizures. History of seizure or condition that may predispose to seizure (including, but not limited to prior cerebrovascular accident, transient ischemic attack, or loss of consciousness within 1 year prior to randomization; brain arteriovenous malformation; or intracranial masses such as a schwannoma or meningioma that is causing edema or mass effect)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Aragon Pharmaceuticals, Inc. Clinical Trial, Study Director — Aragon Pharmaceuticals, Inc.
Locations (12):
- Brazil (6):
  - Ynova Pesquisa Clinica, Florianópolis
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Ensino e Terapia de Inovacao Clinica AMO Etica, Salvador
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo
- Hospital Pablo Tobon Uribe, Medellín, Colombia
- Mexico (5):
  - Instituto Nacional de Cancerologia, México
  - i Can Oncology Center, Monterrey
  - Oncologia Integral Satelite, Naucalpan
  - Centro Oncologico Estatal ISSEMYM, Toluca
  - Farmaco Oncología especializada S.A. de C.V, Zapopan